CLINICAL TRIAL: NCT05378906
Title: A Single-dose, Open-label, Randomized, Crossover Pivotal Bioequivalence Study in Healthy Participants to Assess the Bioequivalence of Darunavir 600 mg in the Presence of Cobicistat 90 mg When Administered as a Fixed Dose Combination Tablet (Darunavir/Cobicistat) Compared to the Co-administration of the Separate Available Formulations (Darunavir 100 mg/mL Suspension at a Dose of 600 mg and Cobicistat 90 mg Tablet), Under Fed Conditions
Brief Title: A Study of Darunavir in the Presence of Cobicistat When Administered as a Fixed Dose Combination Compared to the Co-administration of the Separate Available Formulations of Darunavir and Cobicistat Under Fed Conditions in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR109173; 2021-003955-40 (EudraCT Number); TMC114FD1HTX1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Healthy
MeSH Terms: interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive a single oral dose of darunavir (DRV) and cobicistat (COBI) as one fixed dose combination (FDC) tablet dispersed in water (Treatment A [test]) in Treatment Period 1, followed by a single dose DRV suspension and COBI tablet (Treatment B [Reference]) in Treatment Period 2 on Day 1 of each Treatment Period under fed conditions. There will be a washout period of at least 7 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: DRV/COBI FDC; Drug: COBI; Drug: DRV
- Treatment Sequence BA (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2 on Day 1 of each Treatment Period under fed conditions. There will be a washout period of at least 7 days from dosing on Day 1 of each Treatment Period
  Interventions: Drug: DRV/COBI FDC; Drug: COBI; Drug: DRV

INTERVENTIONS:
Drug: DRV/COBI FDC — Participants will receive a single oral dose of DRV/COBI FDC tablet dispersed in water as per assigned treatment sequence.
  Other Names: TMC114/JNJ-48763364
Drug: COBI — Participants will receive a single oral dose of COBI tablet as per assigned treatment sequence.
  Other Names: JNJ-48763364
Drug: DRV — Participants will receive single oral dose of DRV suspension as per the assigned treatment sequence.
  Other Names: TMC114

SUMMARY:
The purpose of this study is to evaluate the single-dose pharmacokinetic (PK) and bioequivalence of Darunavir (DRV) in the presence of Cobicistat (COBI) when administered as a DRV/COBI fixed dose combination (FDC) tablet dispersed in water compared to the co-administration of the separate available formulations (DRV suspension and COBI tablet) under fed conditions in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening (results must be available on Day -1 of Treatment Period 1). If there are any abnormalities (other than those listed in inclusion criterion 12 [for blood pressure]), they must be considered not clinically relevant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening (results must be available on Day -1 of Treatment Period 1). If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* All women must have a negative highly sensitive serum test (beta-human chorionic gonadotropin [beta-hCG]) 4 days or less before dosing of the first treatment period
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study intervention
* Must sign an informed consent form (ICF) indicating that the participant understands the purpose and procedures required for the study and is willing to participate in the study
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 90 days after last dose

Exclusion Criteria:

* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Clinically significant abnormalities during physical examination, vital signs, or 12-lead ECG at screening or at admission to the study site as deemed appropriate by the investigator
* Known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* With a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillin's, or drug allergy diagnosed in previous studies with experimental drugs
* With a clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Taken any disallowed therapies, concomitant therapy before the planned first dose of study intervention
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Darunavir (DRV) | Pre dose, up to 72 hours post dose (up to Day 4)
  Cmax is defined as the maximum observed plasma concentration of DRV.
Area Under the DRV Concentration-time Curve From Time Zero to Last Quantifiable Time (AUC[0-last]) of DRV | Pre dose, up to 72 hours post dose (up to Day 4)
  AUC (0-last) is the area under the DRV concentration-time curve from time zero to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the DRV Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of DRV | Pre dose, up to 72 hours post dose (up to Day 4)
  AUC (0-infinity) is the area under the DRV concentration-time curve from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z).

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Cobicistat (COBI) | Pre dose, up to 72 hours post dose (up to Day 4)
  Cmax is defined as the maximum observed plasma concentration of COBI.
Area Under the COBI Concentration-time Curve From Time Zero to Last Quantifiable Time (AUC[0-last]) of COBI | Pre dose, up to 72 hours post dose (up to Day 4)
  AUC (0-last) is the area under the COBI concentration-time curve from time zero to the time of the last measurable (non-BQL) concentration, calculated by linear-linear trapezoidal summation.
Area Under the COBI Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of COBI | Pre dose, up to 72 hours post dose (up to Day 4)
  AUC (0-infinity) is the area under the COBI concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z), wherein AUC(0-last) is area under the COBI concentration-time curve from time zero to the time of last measurable non-BQL concentration, C(last) is the last observed measurable (non-BQL) concentration, and lambda(z) is apparent terminal elimination rate constant.
Number of Participants With Serious Adverse Events (SAEs) | Up to 7 weeks
  An SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening (the participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Abnormalities in Physical Examinations | Up to 7 weeks
  Number of participants with abnormalities in physical examinations (including skin examination, body weight, height and family history related to skin disease) will be reported.
Number of Participants with Abnormalities in Vital Sign Measurements | Up to 7 weeks
  Number of participants with abnormalities in vital sign measurements (including temperature, pulse/heart rate, systolic and diastolic blood pressure) will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 7 weeks
  Number of participants with abnormalities in clinical laboratory tests (including hematology, serum chemistry and random urine samples) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Belgium NV, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency